## Relationship and sexual satisfaction of stoma patients

18.04.2022

NCT ID: konstanz\_001

**Information sheet** 

## Questionnaire regarding sexual satisfaction and relationship satisfaction of stoma patients

Thank you very much for participating in an anonymous study regarding sexual and relationship satisfaction of patients with a stoma.

It is the aim of the study to examine sexual and relationship satisfaction of stoma patients. To the best of our knowledge there is no available data regarding this topic. With the results we hope to sensitive health care professionals treating people with a stoma.

The questionnaire is completely anonymous. The data is only accessible by the head of the study and the deputy.

If you have any questions, don't hesitate to contact us.

Dr. Silvan Hämmerli

Head of the study

Phone: 0049 7531 801 1138 silvan.haemmerli@gmail.com

By participating in the study you agree to use the data for publication.

Thank you very much for your time.